CLINICAL TRIAL: NCT00775775
Title: The Relationship Between Fatigue, Sleep Disorders and Endocrine Abnormalities Following Traumatic Brain Injury
Brief Title: Fatigue, Sleep Disorders and Endocrine Abnormalities in TBI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Anthony Lequerica, Ph.D., Kessler Foundation Research Center
Other Study IDs: R45303
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TBI: Patients with moderate to severe TBI

SUMMARY:
This study will test if patients with moderate to severe traumatic brain injuries also have endocrine abnormalities, examine any existing relationships among fatigue, depression and endocrine abnormalities, and the relationship between endocrine abnormalities, quality of life, and community integration.

ELIGIBILITY:
Inclusion Criteria:

* Having moderate to severe TBI at least 3 months prior to enrollment. This can be demonstrated by a history of loss of consciousness, amnesia or another neurologic deficit after brain injury
* Be between the ages of 18 and 70 years

Exclusion Criteria:

* History of prior TBI, stroke, seizures, severe psychiatric disturbances (i.e., those known to influence memory performance, such as schizophrenia, bipolar disorder), or drug abuse will be excluded.
* Pregnant, nursing, or planning pregnancy during the study period.
* Dementia
* Other neurological conditions which are associated with aging and known to cause fatigue (e.g. Parkinson's Disease)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of 50 participants taken from the outpatient brain injury program at Kessler.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2003-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To further study the incidence of fatigue and endocrine abnormalities in an outpatient TBI population | 1 year

SECONDARY OUTCOMES:
To study the relationship between fatigue and endocrine abnormalities | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lequerica, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States